CLINICAL TRIAL: NCT02878356
Title: Acquisition of MI Competence Trough the Training Methods Used in the Swedish County Councils and Municipalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Ministry of Health and Social Affairs, Sweden (Other Government)
Responsible Party: Principal Investigator, Lars Forsberg, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R30024-2 AAMR
Record Dates: First submitted 2014-02-13; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Competence
Keywords: Motivational Interviewing, Clinical supervision, Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regular MI-training (Active Comparator): Regular training (n= 59) the Motivational Interviewing (MI) -training methods used in the Swedish county councils and municipalities
  Interventions: Behavioral: Regular MI-training
- Regular MI-training + supervision half (Active Comparator): Regular MI-training followed by six individual MI-supervision sessions at monthly intervals based on only the behavior counts component of MITI (n= 58)
  Interventions: Behavioral: Regular MI-training; Behavioral: Regular MI-training + supervision half
- Regular MI-training + supervision full (Active Comparator): Regular MI-training followed by MI-supervision based on both the behavior counts and the five global dimensions of MITI (n= 58)
  Interventions: Behavioral: Regular MI-training; Behavioral: Regular MI-training + supervision full

INTERVENTIONS:
Behavioral: Regular MI-training — Regular training (n= 59) the Motivational Interviewing (MI) -training methods used in the Swedish county councils and municipalities
Behavioral: Regular MI-training + supervision half — Regular MI-training followed by six individual MI-supervision sessions at monthly intervals based on only the behavior counts component of MITI (n= 58)
  Arms: Regular MI-training + supervision half
Behavioral: Regular MI-training + supervision full — Regular MI-training followed by MI-supervision based on both the behavior counts and the five global dimensions of MITI (n= 58)
  Arms: Regular MI-training + supervision full

SUMMARY:
In the Swedish county councils and municipalities, Motivational Interviewing (MI) training with different forms and content is taking place as part of the implementation of the method. The study aims to evaluate to what extent the practitioners acquire and retain MI skills trough the different training methods used by comparing them with a format that in previous studies has shown to be required for the long-term acquisition of proficiency in MI; training including supervision consisting of feedback based on monitoring of practice.

DETAILED DESCRIPTION:
The basis for a successful implementation of an evidence-based treatment in routine clinical care is quality assessment of all stages of delivery, implementation and evaluation. In the Swedish county councils and municipalities, Motivational Interviewing (MI) training with different forms and content is taking place as part of the implementation of the method.

Aims: To evaluate to what extent the practitioners acquire and retain MI skills through the different training methods used in the Swedish county councils and municipalities by comparing them with a format that in previous studies has shown to be required for the long-term acquisition of proficiency in MI; training including supervision consisting of feedback based on monitoring of practice.

Method: In 2013-2014, 175 practitioners that attend MI training in five different county councils and municipalities in Sweden will be randomized to one of the study's three groups: (a) "Regular training" (n= 66), b) "Regular training" followed by six individual supervision sessions at monthly intervals based on only the behavior counts component of the Motivational Interviewing Treatment Integrity (MITI) Code (n= 67), and (c) "Regular training" followed by supervision based on both the behavior counts and the five global dimensions of the MITI (n= 67). All practitioners will record three sessions: one before " regular training", one after "regular training" and one six month after training. The practitioners in group b and c will record five additional sessions in conjunction with the supervision. All supervision and recording sessions will be made over the phone with actors role-playing clients. The sessions will be assessed for proficiency in MI by MIC Lab at the Karolinska Institute according to the Swedish translation of MITI 3.1.

Time Frame: The specific time points at which the outcome measure (the Swedish version of the MITI, version 3.1.) will be assessed are:

1. Before the county councils' workshop trainings (pre-workshop).
2. Directly after the workshop trainings (post-workshop).
3. Six months after the workshop trainings (follow-up). => Since the different county council workshop trainings differ in time (e.g. one to four month) the participants from the different county councils will be followed for a period in between seven month (one + six) to ten month (four + six).

The participants randomized to the two groups with additional supervision will also be assessed five times between the post-workshop and the follow-up assessment (e.g. every month).

ELIGIBILITY:
Inclusion Criteria:

• Subjects are practitioners that attend MI-training in five different Swedish county councils 2013-2014.

Exclusion Criteria:

• Practitioners younger than 18 and older than 65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Acquisition of MI competence | Change from Baseline (pre-workshop) in MI competence assessed by the Swedish version of the MITI, directly after the workshop trainings (post-workshop), and six months after the workshop trainings (follow-up).
  The effectiveness of the county council workshop trainings will be measured with mean differences between the pre- and post-workshop assessment. The impact of the additional telephone supervision on the county councils' workshop trainings will be measured with mean differences between the post-workshop and the follow-up assessment.
  All acquisition of MI competence will be assessed by the Swedish version of the MITI, version 3.1. The MITI is a coding system with good psychometric properties widely used as a treatment integrity measure and as a feedback tool to improve MI skills in training and in clinical practice (Moyers, Martin, Manuel, Hendrickson, & Miller: Assessing competence in the use of motivational interviewing. Journal of Substance Abuse Treatment 2005, 28:19-26.).

CONTACTS AND LOCATIONS:
Overall Officials: Lars Forsberg, PhD, Study Director — Karolinska Institutet
Locations (1):
- MIC Lab, Department of Clinical Neuroscience, Karolinska Institutet, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available.